CLINICAL TRIAL: NCT06628154
Title: The Effects of Single-dose Losartan on Cognitive Flexibility and Learning in Healthy Adults: a Randomised Controlled Study
Brief Title: Losartan and Emotional Learning
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford Health Biomedical Research Centre (OH BRC) support scheme (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R80447
Record Dates: First submitted 2024-09-30; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Emotional Processing
Keywords: emotional processing; reward; anxiety; depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: Parallel randomised experimental medicine trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- losartan (Experimental): oral single-dose losartan potassium (Cozaar; 50mg)
  Interventions: Drug: Losartan potassium 50mg
- placebo (Placebo Comparator): Microcellulose placebo in identical capsule
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Losartan potassium 50mg — Single dose losartan (50 mg, weight-adjusted), encapsulated identically to placebo
  Arms: losartan
Other: Placebo — Single tablet encapsulated identically to losartan
  Arms: placebo

SUMMARY:
This study explores the effects of single-dose losartan (50mg) versus placebo on emotional processing in healthy volunteers.

DETAILED DESCRIPTION:
The renin-angiotensin system is a major hormone system involved in blood pressure regulation. However, its major receptors are also found in the brain, particularly in areas implicated in anxiety and depression. In line with this topography, drugs blocking angiotensin-II receptors have been shown to have effects on cognition that are opposite to those seen in emotional disorders. For instance, angiotensin receptor blockade improves fear extinction, and it dampens stress responsivity to highly aversive images. In line with such cognitive effects, population-based studies suggest that angiotensin receptor blockers - compared to other antihypertensive drugs - prevent the development of post-traumatic stress disorder following trauma exposition and improve outcomes in patients taking SSRI.

This study aims to shed further light on how the renin-angiotensin system affects different aspects of cognitive processing in humans relevant to emotional disorders. In a double-blind, randomized between-group design, we will investigate the effects of a single dose of losartan (50mg) versus placebo on emotional processing in N=60 healthy volunteers aged 18-50 years. Results from this study will help us understand how the renin-angiotensin system affects emotional processing in humans, and they will help us identify potential synergistic overlaps with the cognitive mechanisms of action of effective treatment of emotional disorders.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Aged 18-50 years
* Score of or below 45 on the Dimensional Anhedonia Rating Scale (DARS; Rizvi et al., 2015)
* Sufficient written and spoken English skills to understand what the study involves, and to complete the questionnaires
* Non- or light-smoker (5 cigarettes a day)

Exclusion Criteria:

* Past or present DSM-5 axis-I diagnosis (based on SCID results at screening) other than anxiety disorder, dysthymia or unipolar depression
* First-degree family member with severe psychiatric illness
* CNS-medication last 6 weeks (including as part of another study)
* Current blood pressure or other heart medication (especially aliskiren or beta blockers)
* Diagnosis of intravascular fluid depletion or dehydration
* History of angioedema
* Impaired kidney function (based on self-report)
* Very low blood pressure (defined as repeated (at least three consecutive measurements) measures of blood pressure under standardised conditions where either the systolic or the diastolic blood pressure or both are below 90/50 mmHg (in accordance with established standard definitions: DOI 10.1186/s12887-016-0633-7))
* Lifetime history of epilepsy or other neurological disease (e.g. autism, ADHD)
* Lifetime history of systemic infection, or clinically significant hepatic, cardiac, obstructive respiratory, renal, cerebrovascular, metabolic, endocrine or pulmonary disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study
* Significant loss of hearing that is not corrected with a hearing device
* Women: pregnancy, breast-feeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Reinforcement Learning | 1 hour after capsule intake
  reinforcement learning, calculated as the learning rate from aversive and appetitive decision outcomes. Larger scores indicate better learning from an outcome.

SECONDARY OUTCOMES:
Cognitive Flexibility | 1 hour after capsule intake
  switch cost, calculated by rank-ordering the differences between each switch trial RT and each participants average RT for all non-switch trials from 1 - 10 (with better and worse bins having values closer to 1 and 10, respectively), and then summing the bin values to compute a total bin score for each participant. Inaccurate responses are penalized by being assigned a score of 20. Smaller bin scores indicate greater accuracy and lower RT.
AAT effect score | 1hour after capsule intake
  mean reaction time of the pull trials of a valence category subtracted from the push trials of the same category, yielding a single indicator of approach/avoidance, with positive scores indicating relatively stronger approach and negative scores indicating relatively stronger avoidance
Motivational effort in the Apples Task | 1hour after capsule intake
  effort valuation, calculated as the willingness to engage in physical effort to obtain rewards of certain values using the Apples Task (and computational approaches)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Reinecke, PhD, Principal Investigator — University of Oxford
Locations (1):
- Warneford Hospital, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided